CLINICAL TRIAL: NCT01718353
Title: Phase II Trial to Evaluate Benefit of Early Switch From First-Line Docetaxel/Prednisone to Cabazitaxel/Prednisone and the Opposite Sequence, Exploring Molecular Markers and Mechanisms of Taxane Resistance in Men With Metastatic Castration-Resistant Prostate Cancer (mCRPC) Who Have Not Received Prior Chemotherapy
Brief Title: Early Switch From First-Line Docetaxel/Prednisone to Cabazitaxel/Prednisone and the Opposite Sequence, Exploring Molecular Markers in Men With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Acronym: TAXYNERGY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABAZL06056; U1111-1130-9893 (Other: UTN)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2016-08

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — Docetaxel; cabazitaxel; XRP6258; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel + Prednisone (Treatment A) (Experimental): Docetaxel 75 mg/m^2 intravenous (IV) infusion on Day 1 of Cycle 1 and every 3 weeks (q3w) thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily. Participants with <30% PSA reduction from baseline at the end of Cycle 4 switched to Cabazitaxel 25mg/m^2 IV infusion on Day 1 of Cycle 5 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily until disease progression (DP), death, unacceptable toxicity or participant's refusal of further study treatment. Participants with ≥30% PSA reduction from baseline at the end of Cycle 4, continued on the same treatment which they received before switching until DP, death, unacceptable toxicity or participant's refusal of further study treatment.
  Interventions: Drug: DOCETAXEL (XRP6976); Drug: Prednisone
- Cabazitaxel + Prednisone (Treatment B) (Experimental): Cabazitaxel 25 mg/m^2 IV infusion on Day 1 of Cycle 1 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily. Participants with <30% PSA reduction from baseline at the end of Cycle 4 switched to Docetaxel 75mg/m^2 IV infusion on Day 1 of Cycle 5 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily until DP, death, unacceptable toxicity or participant's refusal of further study treatment. Participants with ≥30% PSA reduction from baseline at the end of Cycle 4, continued on the same treatment which they received before switching until DP, death, unacceptable toxicity or participant's refusal of further study treatment.
  Interventions: Drug: CABAZITAXEL (XRP6258); Drug: Prednisone

INTERVENTIONS:
Drug: DOCETAXEL (XRP6976) — Pharmaceutical form: Concentrate for solution for infusion Route of administration: Intravenous
  Other Names: Taxotere®
  Arms: Docetaxel + Prednisone (Treatment A)
Drug: CABAZITAXEL (XRP6258) — Pharmaceutical form: Concentrate and solvent for solution for infusion Route of administration: Intravenous
  Other Names: Jevtana®
  Arms: Cabazitaxel + Prednisone (Treatment B)
Drug: Prednisone — Pharmaceutical form: Tablet Route of administration: Oral

SUMMARY:
Docetaxel and cabazitaxel are cancer chemotherapy agents of the taxane drug class. The purpose of this study is to explore the benefit, for treatment of metastatic castration-resistant prostate cancer (mCRPC), of a regimen in which participants begin treatment with either of these two taxane drugs (docetaxel or cabazitaxel, in combination with prednisone) and are switched to the other taxane drug if prostate-specific antigen (PSA) value does not decrease ≥30% after 4 cycles. As defined in study protocol amendment 3, efficacy results are summarized for all participants combined, irrespective of which agent (docetaxel or cabazitaxel) was administered initially, rather than separately for the two groups based on taxane administered initially. One of the primary outcome measures is percentage of participants with a ≥50% sustained decrease from baseline in PSA at any time during the trial. By providing an opportunity for patients to switch taxane based on early PSA response, there may be a difference in result for this measure versus result in a study where it was not possible to switch. The other primary outcome measures are change from baseline in circulating tumor cells (CTCs) biomarkers percent androgen receptor nuclear localization (%ARNL) and microtubule bundling (MTB).

DETAILED DESCRIPTION:
* Participants were treated until progressive disease, unacceptable toxicity, death, or participant's refusal of further study treatment. All participants were followed until death or the study cut-off date, whichever came first.
* Study cut-off was 1 month after the last participant last treatment.
* Participants alive at the cut-off date were not followed for overall survival.

ELIGIBILITY:
Inclusion criteria :

* Histologically- or cytologically-confirmed prostate adenocarcinoma with documented distant metastases (M1 disease).
* Progressive disease while receiving hormonal therapy or after surgical castration.
* Effective castration (serum testosterone levels ≤50 ng/dL) by orchiectomy and/or luteinizing hormone releasing hormone agonists or antagonist with or without anti-androgens.

Exclusion criteria:

* Prior chemotherapy for prostate cancer, except estramustine and adjuvant/neoadjuvant treatment completed >3 years ago. Prior treatment with sipuleucel-T immunotherapy was allowed at the condition participant did not receive prior chemotherapy.
* Less than 28 days elapsed from prior treatment with estramustine, radiotherapy or surgery to the time of random allocation.
* Prior beta isotope therapy, whole pelvic radiotherapy, or radiotherapy to >30% of bone marrow.
* Adverse events (excluding alopecia and those listed in the specific exclusion criteria) from any prior anticancer therapy of grade >1(National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v4.03) at the time of random allocation.
* Less than 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status >2.
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
* Prior malignancy. Adequately treated basal cell or squamous cell skin or superficial (pTis, pTa and pT1) bladder cancer were allowed, as well as any other cancer for which chemotherapy had been completed ≥3 years ago and from which the participant had been disease-free for ≥3 years.
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to random allocation.
* Any of the following within 6 months prior to study enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III or IV congestive heart failure, stroke or transient ischemic attack.
* Any of the following within 3 months prior to random allocation: treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism, or other uncontrolled thromboembolic event.
* Acquired immunodeficiency syndrome (AIDS)-related illnesses or known HIV disease requiring antiretroviral treatment.
* Any severe acute or chronic medical condition which could impair the ability of the participant to participate in to the study or interfere with interpretation of study results, or participant unable to comply with the study procedures.
* Concomitant treatment with biphosphonates or denosumab except if the dose had been stable for 4 weeks prior to enrollment.
* Absence of signed and dated Institutional Review Board (IRB)-approved participant informed consent prior to enrollment into the study.
* Participants with reproductive potential who did not agree to use an accepted and effective method of contraception during the study treatment period. The definition of "effective method of contraception" was based on the investigator's judgment.
* History of hypersensitivity to docetaxel or polysorbate 80.
* Inadequate organ and bone marrow function.
* Contraindications to the use of corticosteroid treatment.
* Symptomatic peripheral neuropathy grade >2 (NCI CTCAE v.4.03).
* Treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a two-week wash-out period was necessary for participants who were already on these treatments).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (19):
- United States (14):
  - Investigational Site Number 840003, Birmingham, Alabama
  - Investigational Site Number 840102, Washington D.C., District of Columbia
  - Investigational Site Number 840005, Indianapolis, Indiana
  - Investigational Site Number 840025, Metairie, Louisiana
  - Investigational Site Number 840002, Baltimore, Maryland
  - Investigational Site Number 840007, Bethesda, Maryland
  - Investigational Site Number 840017, Rockville, Maryland
  - Investigational Site Number 840010, Cherry Hill, New Jersey
  - Investigational Site Number 840015, East Orange, New Jersey
  - Investigational Site Number 840001, New York, New York
  - Investigational Site Number 840013, New York, New York
  - Investigational Site Number 840009, Charleston, South Carolina
  - Investigational Site Number 840012, Seattle, Washington
  - Investigational Site Number 840004, Madison, Wisconsin
- Canada (5):
  - Investigational Site Number 124001, Edmonton, Alberta
  - Investigational Site Number 124004, Montreal, Quebec
  - Investigational Site Number 124002, Montreal, Quebec
  - Investigational Site Number 124006, Québec, Quebec
  - Investigational Site Number 124005, Sherbrooke, Quebec

REFERENCES:
- [Derived] Tagawa ST, Antonarakis ES, Gjyrezi A, Galletti G, Kim S, Worroll D, Stewart J, Zaher A, Szatrowski TP, Ballman KV, Kita K, Tasaki S, Bai Y, Portella L, Kirby BJ, Saad F, Eisenberger MA, Nanus DM, Giannakakou P. Expression of AR-V7 and ARv567es in Circulating Tumor Cells Correlates with Outcomes to Taxane Therapy in Men with Metastatic Prostate Cancer Treated in TAXYNERGY. Clin Cancer Res. 2019 Mar 15;25(6):1880-1888. doi: 10.1158/1078-0432.CCR-18-0320. Epub 2018 Oct 9. PMID 30301829
- [Derived] Antonarakis ES, Tagawa ST, Galletti G, Worroll D, Ballman K, Vanhuyse M, Sonpavde G, North S, Albany C, Tsao CK, Stewart J, Zaher A, Szatrowski T, Zhou W, Gjyrezi A, Tasaki S, Portella L, Bai Y, Lannin TB, Suri S, Gruber CN, Pratt ED, Kirby BJ, Eisenberger MA, Nanus DM, Saad F, Giannakakou P; TAXYNERGY Investigators. Randomized, Noncomparative, Phase II Trial of Early Switch From Docetaxel to Cabazitaxel or Vice Versa, With Integrated Biomarker Analysis, in Men With Chemotherapy-Naive, Metastatic, Castration-Resistant Prostate Cancer. J Clin Oncol. 2017 Oct 1;35(28):3181-3188. doi: 10.1200/JCO.2017.72.4138. Epub 2017 Jun 20. PMID 28632486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 centers in Canada and United States. A total of 81 participants were screened between 20 March 2013 and 29 May 2014, of which, 63 participants were randomized and 61 were treated. A total of 18 participants were screen failure mainly due to exclusion criteria met and inclusion criteria not met.
Pre-assignment Details: Participants were randomized by Interactive Voice Response System (IVRS) in 2:1 ratio (Treatment A : Treatment B) to receive either Treatment A (Docetaxel + Prednisone) or Treatment B (Cabazitaxel + Prednisone).
Groups:
- Docetaxel + Prednisone (Treatment A): Docetaxel 75 mg/m^2 intravenous (IV) infusion on Day 1 of Cycle 1 and every 3 weeks (q3w) thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily. Participants with <30% prostate-specific antigen (PSA) reduction from baseline at the end of Cycle 4 switched to Cabazitaxel 25mg/m^2 IV infusion on Day 1 of Cycle 5 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily until disease progression (DP), death, unacceptable toxicity or participant's refusal of further study treatment. Participants with ≥30% PSA reduction from baseline at the end of Cycle 4, continued on the same treatment which they received before switching until DP, death, unacceptable toxicity or participant's refusal of further study treatment.
Period: Overall Study
Arm/Group | Docetaxel + Prednisone (Treatment A) | Cabazitaxel + Prednisone (Treatment B)
Started | 41 | 22
Treated | 39 | 22
Treated up to End of Cycle 4 | 32 (7 participants discontinued before Cycle 5) | 16 (6 participants discontinued before Cycle 5)
Treated From Cycle 5 | 23 (12 participants switched from Treatment A to B & 3 participants switched from Treatment B to A.) | 25 (3 participants switched from Treatment B to A & 12 participants switched from Treatment A to B.)
Completed | 29 (Participants at study cut-off, Adverse Event (AE), DP & consent withdrawn were considered completed.) | 17 (Participants at study cut-off, AE, DP and consent withdrawn were considered completed.)
Not Completed | 12 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Principal Investigator's Decision | 10 | 4
Not completed — Randomized but not treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel + Prednisone (Treatment A): Docetaxel 75 mg/m^2 IV infusion on Day 1 of Cycle 1 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily. Participants with <30% PSA reduction from baseline at the end of Cycle 4 switched to Cabazitaxel 25mg/m^2 IV infusion on Day 1 of Cycle 5 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily until DP, death, unacceptable toxicity or participant's refusal of further study treatment. Participants with ≥30% PSA reduction from baseline at the end of Cycle 4, continued on the same treatment which they received before switching until DP, death, unacceptable toxicity or participant's refusal of further study treatment.
- Total: Total of all reporting groups
Arm/Group | Docetaxel + Prednisone (Treatment A) | Cabazitaxel + Prednisone (Treatment B) | Total
Number analyzed (Participants) | 41 | 22 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (7.8) | 69.2 (9.5) | 69.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 22 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With PSA Response
Description: PSA response was defined as ≥50% decrease in PSA levels in both treatment arms from baseline, during the whole treatment, before treatment switch and after treatment switch. PSA progression was defined as decline of PSA from baseline (an increase of ≥25% [at least 2ng/ml] over the nadir value, confirmed by a second PSA value at least 3 weeks apart) and no decline of PSA from baseline (an increase of ≥25% [at least 2ng/ml] over the baseline value after 12 weeks of treatment, confirmed by a second PSA value at least 3 weeks apart). Because the purpose of this study is to explore the benefit of a regimen in which participants are switched to a different taxane if PSA does not decrease ≥30% after 4 cycles, irrespective of which agent (docetaxel or cabazitaxel) is administered initially, the data for participants who began treatment with docetaxel and for those who began treatment with cabazitaxel were combined for the efficacy analyses.
Time Frame: Baseline, Pre-dose every 3 weeks, 30 days after last treatment administration (End of treatment [EOT]), every 3 months (for 1 year) then every 6 months until PSA progression or study cut-off, whichever was earlier (Maximum duration: 60 weeks)
Population: Analysis was performed on all randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- Overall Population (Treatment A or Treatment B): Docetaxel 75 mg/m^2 or Cabazitaxel 25 mg/m^2 IV infusion on Day 1 of Cycle 1 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily. Participants with <30% PSA reduction from baseline at the end of Cycle 4, switched to Cabazitaxel 25 mg/m^2 IV or Docetaxel 75mg/m^2 IV infusion respectively on Day 1 of Cycle 5 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily until DP, death, unacceptable toxicity or participant's refusal of further study treatment. Participants with ≥30% PSA reduction from baseline at the end of Cycle 4, continued on the same treatment which they received before switching until DP, death, unacceptable toxicity or participant's refusal of further study treatment.
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 63
percentage of participants
  PSA response before switch | 39.7
  PSA response after switch | 15.9
  Overall PSA response | 55.6

2. Primary Outcome: Drug-target Engagement in Circulating Tumor Cells (CTCs): Change From Baseline at Cycle 1 Day 8 in Percent Androgen Receptor Nuclear Localization (%ARNL) by Categories of PSA Decrease From Baseline (≥50%, Not ≥50%) After Cycle 4
Description: Analysis of CTCs is a co-primary endpoint. Growth of prostate cancer cells is dependent on sustained androgen receptor (AR) nuclear signaling. Taxanes (e.g., docetaxel and cabazitaxel) may mediate some of their activity in prostate cancer by impairing AR trafficking along the microtubules from the tumor cell cytoplasm into the nucleus, as a result of taxane-induced microtubule bundling (MTB). Blood samples were collected at baseline and post-treatment to allow isolation of CTCs, which were evaluated for tumor cell biomarker measures %ARNL and MTB score. %ARNL was assessed by quantitative analysis of images of CTCs captured by geometrically enhanced differential immunocapture (GEDI). Reduction from baseline in %ARNL (percentage of total cellular AR that is located in the nucleus) may indicate inhibition of AR signaling. Change from baseline in %ARNL at Cycle 1 Day 8 is summarized by categories of participants with PSA decrease from baseline (≥50%, Not ≥50%) after Cycle 4.
Time Frame: Baseline and Cycle 1 Day 8, Cycle 4
Population: Participants with evaluable CTCs at both baseline and Cycle 1 Day 8, and evaluable PSA result at both baseline and Cycle 4
Measure: Mean (Standard Deviation); unit: percentage ARNL
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 19
percentage ARNL
  PSA decreased ≥50% at Cycle 4: number analyzed (Participants) | 9
  PSA decreased ≥50% at Cycle 4 | -17.58 (21.54)
  PSA not decreased ≥50% at Cycle 4: number analyzed (Participants) | 10
  PSA not decreased ≥50% at Cycle 4 | 2.30 (11.16)
Statistical Analysis 1: Comparison: Overall Population (Treatment A or Treatment B); %ARNL change from baseline at Cycle 1 Day 8 in participants with ≥50% decrease in PSA at Cycle 4 was compared with that of participants who did not have ≥50% decrease in PSA at Cycle 4; Test type: Other; p = 0.02, ANOVA

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval between the date of random allocation of the treatment and the date of first documentation of any of the following: radiographic tumor progression (using Modified Response Evaluation Criteria in Solid Tumors [RECIST1.1] before any switch and during the study), clinical progression (including skeletal-related events, increasing pain requiring escalation of narcotic analgesics, urinary obstruction), PSA progression or death from any cause. Analysis was performed by Kaplan Meier method.
Time Frame: From Baseline until DP or death due to any cause or study cut off, whichever was earlier (Maximum duration: 60 weeks)
Population: Analysis was performed on all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 63
months
  Before switch | 4.1 [3.81 to NA] — The upper bound of the confidence interval could not be estimated because of insufficient number of events for before switch PFS.
  Whole treatment continuum | 9.1 [4.93 to 11.70]

4. Secondary Outcome: PSA Progression Free Survival
Description: PSA progression-free survival before any switch and PSA progression free survival during the study was defined as the time interval between the date of Day 1 of Cycle 1 to the date of either first PSA progression or death due to any cause whichever came first. PSA progression was defined as decline of PSA from baseline (an increase of ≥25% [at least 2ng/mL] over the nadir value, confirmed by a second PSA value at least 3 weeks apart) and no decline of PSA from baseline (an increase of ≥25% [at least 2ng/mL] over the baseline value after 12 weeks of treatment, confirmed by a second PSA value at least 3 weeks apart).
Time Frame: From Baseline until DP or death due to any cause or study cut off date, whichever was earlier (Maximum duration: 60 weeks)
Population: Analysis was performed on all randomized population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 63
months
  Before switch | NA [3.09 to NA] — The median and upper bound of the confidence interval could not be estimated because of insufficient number of events for before switch PSA PFS.
  whole treatment continuum | 12.4 [8.31 to NA] — The upper bound of the confidence interval could not be estimated because of insufficient number of events for whole treatment continuum PSA PFS.

5. Secondary Outcome: Percentage of Participants With Objective Response
Time Frame: From baseline until DP or study cut off, whichever was earlier (Maximum duration: 60 weeks)
Population: No data was collected to determine the Objective Response, hence this outcome measure was not evaluated.
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 0

6. Secondary Outcome: Radiographic Progression-free Survival (rPFS)
Time Frame: From baseline, every 12 weeks until radiological tumor progression or study cut-off, whichever was earlier (Maximum duration: 60 weeks)
Population: Analysis was performed on all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 63
months | NA [NA to NA] — Kaplan-Meier was not analyzed, as less than 50% population had the event. Hence, data was not calculated and reported.

7. Secondary Outcome: Clinical Progression-free Survival (cPFS)
Description: cPFS was assessed before switch and during the study including skeletal-related events (SRE), increasing pain requiring escalation of narcotic analgesics, urinary obstruction, etc. SRE included pathological fractures and/or spinal cord compression, need for bone irradiation (including radioisotopes or bone surgery), change of antineoplastic therapy (including introduction of bisphosphonates or denosumab in the face of increase in pain) to treat bone pain. Pain was assessed using present pain intensity (PPI) scale (0=no pain, up to 5=excruciating pain) and analgesics used for cancer pain (1 point for non-narcotic medications and 4 points for narcotic medications).
Time Frame: Baseline, Pre-dose every 3 weeks, EOT, every 3 months (for 1 year) until first SRE occurrence or death or study cut-off, whichever was earlier (Maximum duration: 60 weeks)
Population: Analysis was performed on all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 63
months
  Before switch | NA [7.16 to NA] — The median and upper bound of the confidence interval could not be estimated because of insufficient number of events for before switch cPFS.
  Whole treatment continuum | NA [NA to NA] — Kaplan-Meier was not analyzed, as less than 50% population had the event. Hence, data was not calculated and reported.

8. Secondary Outcome: Overall Survival
Description: Overall survival before switch and overall survival during the study was defined as the time interval from the date of random allocation to the date of death due to any cause until study cut-off date.
Time Frame: From baseline until death due to any cause or study cut-off, whichever was earlier (Maximum duration: 60 weeks)
Population: Analysis was performed on all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 63
Months
  Before switch | 8.8 [4.01 to NA] — Not enough events were reported to calculate Kaplan-Meier curve.
  whole treatment continuum | NA [14.03 to NA] — Not enough events were reported to calculate Kaplan-Meier curve.

9. Secondary Outcome: Percentage of Participants With ≥30% and ≥50% Reduction in PSA Response
Description: Participants with ≥30% and ≥50% reduction in PSA response from base line were evaluated in participants who were previously treated with a high potency androgen receptor (AR)-targeted agent (AR signaling inhibitor or cytochrome P450 17 alphahydroxylase/17,20lyase [CYP 17] inhibitor).
Time Frame: From baseline until DP or study cut-off, whichever was earlier (Maximum duration: 60 weeks)
Population: Analysis was performed on as-treated population that included all participants who received initial taxane treatment and had a post treatment assessment. Number of participants analyzed=participants treated/non-treated with AR-target agent and with PSA response assessment at specified time-points.
Measure: Number; unit: percentage of participants
Groups:
- Overall Population (AR-target Agent Treated): Participants having prior treatment experience with a high potency AR targeted agent (AR signaling inhibitor or CYP 17) before this study.
- Overall Population (Non AR-target Agent Treated): Participants not having prior treatment experience with a high potency AR targeted agent (AR signaling inhibitor or CYP 17 inhibitor) before this study.
Arm/Group | Overall Population (AR-target Agent Treated) | Overall Population (Non AR-target Agent Treated)
Number analyzed (Participants) | 25 | 35
percentage of participants
  ≥30% reduction | 52.0 | 74.3
  ≥50% reduction | 44.0 | 68.6

10. Primary Outcome: Drug-target Engagement in CTCs: Change From Baseline at Cycle 1 Day 8 in MTB by Categories of PSA Decrease From Baseline (≥30%, Not ≥30%) After Cycle 4
Description: Analysis of CTCs is a co-primary endpoint. Growth of prostate cancer cells is dependent on sustained AR nuclear signaling. Taxanes (e.g., docetaxel and cabazitaxel) may mediate some of their activity in prostate cancer by impairing AR trafficking along the microtubules from the tumor cell cytoplasm into the nucleus, as a result of taxane-induced MTB. Blood samples were collected at baseline and post-treatment to allow isolation of CTCs, which were evaluated for tumor cell biomarker measures %ARNL and MTB score. MTB in images of CTCs captured by GEDI was qualitatively assessed by three independent operators for increase compared with baseline on a scale of 0 to 3 from no to most MTB increase. Increase from baseline in MTB may indicate inhibition of AR signaling. Change from baseline in MTB at Cycle 1 Day 8 is summarized by categories of participants with PSA decrease from baseline (≥30%, Not ≥30%) after Cycle 4.
Time Frame: Baseline and Cycle 1 Day 8, Cycle 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Population (Treatment A or Treatment B)
Number analyzed (Participants) | 19
units on a scale
  PSA decreased ≥30% at Cycle 4: number analyzed (Participants) | 12
  PSA decreased ≥30% at Cycle 4 | 0.69 (0.87)
  PSA not decreased ≥30% at Cycle 4: number analyzed (Participants) | 7
  PSA not decreased ≥30% at Cycle 4 | 0.09 (0.18)
Statistical Analysis 1: Comparison: Overall Population (Treatment A or Treatment B); MTB change from baseline at Cycle 1 Day 8 in participants with ≥30% decrease in PSA at Cycle 4 was compared with that of participants who did not have ≥30% decrease in PSA at Cycle 4; Test type: Other; p = 0.0927, ANOVA

ADVERSE EVENTS:
Description: Reported AEs are treatment emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the time of first dose until 30 days after the last treatment administration). Safety population includes all treated participants.
Groups:
- Docetaxel + Prednisone (Treatment A) - Throughout: Docetaxel 75 mg/m^2 IV infusion on Day 1 of Cycle 1 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily. Participants with ≥30% PSA reduction from baseline at the end of Cycle 4, continued on the same treatment throughout until DP, death, unacceptable toxicity or participant's refusal of further study treatment.
- Cabazitaxel + Prednisone (Treatment B) - Throughout: Cabazitaxel 25 mg/m^2 IV infusion on Day 1 of Cycle 1 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily. Participants with ≥30% PSA reduction from baseline at the end of Cycle 4, continued on the same treatment throughout until DP, death, unacceptable toxicity or participant's refusal of further study treatment.
- Switched Population (Treatment A to B or Treatment B to A): Docetaxel 75 mg/m^2 or Cabazitaxel 25 mg/m^2 IV infusion on Day 1 of Cycle 1 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily. Participants with <30% PSA reduction from baseline at the end of Cycle 4 switched to Cabazitaxel 25 mg/m^2 IV or Docetaxel 75mg/m^2 IV infusion respectively on Day 1 of Cycle 5 and q3w thereafter, in combination with Prednisone (or Prednisolone) 10 mg orally daily until DP, death, unacceptable toxicity or participant's refusal of further study treatment.
Arm/Group | Docetaxel + Prednisone (Treatment A) - Throughout | Cabazitaxel + Prednisone (Treatment B) - Throughout | Switched Population (Treatment A to B or Treatment B to A)
Serious Adverse Events (participants affected / at risk) | 10/27 | 8/19 | 9/15
Other Adverse Events (participants affected / at risk) | 26/27 | 18/19 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Prednisone (Treatment A) - Throughout (N=27) | Cabazitaxel + Prednisone (Treatment B) - Throughout (N=19) | Switched Population (Treatment A to B or Treatment B to A) (N=15)
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaphylactoid reaction (Immune system disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1
Nerve root compression (Nervous system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Prednisone (Treatment A) - Throughout (N=27) | Cabazitaxel + Prednisone (Treatment B) - Throughout (N=19) | Switched Population (Treatment A to B or Treatment B to A) (N=15)
Urinary tract infection (Infections and infestations) | 1 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic phlebitis (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 2 | 3
Agitation (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 9 | 6 | 3
Dizziness (Nervous system disorders) | 3 | 3 | 3
Dysgeusia (Nervous system disorders) | 4 | 2 | 3
Paraesthesia (Nervous system disorders) | 3 | 2 | 3
Headache (Nervous system disorders) | 3 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 5 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 2 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 3 | 2 | 0
Flushing (Vascular disorders) | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 1 | 1
Hot flush (Vascular disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 12 | 9
Nausea (Gastrointestinal disorders) | 8 | 10 | 7
Abdominal pain (Gastrointestinal disorders) | 7 | 4 | 4
Constipation (Gastrointestinal disorders) | 3 | 6 | 5
Vomiting (Gastrointestinal disorders) | 3 | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 3 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 5 | 5
Nail ridging (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 5
Dysuria (Renal and urinary disorders) | 1 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1
Fatigue (General disorders) | 18 | 13 | 10
Oedema peripheral (General disorders) | 7 | 3 | 4
Pyrexia (General disorders) | 3 | 2 | 1
Asthenia (General disorders) | 3 | 0 | 1
Hyperthermia (General disorders) | 3 | 0 | 0
Chills (General disorders) | 2 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 3 | 1
Blood creatinine increased (Investigations) | 1 | 2 | 0
Weight increased (Investigations) | 2 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.